CLINICAL TRIAL: NCT00149422
Title: Can Pro-brain-natriuretic Peptide Guided Therapy of Chronic Heart Failure Improve Heart Failure Morbidity and Mortality?
Brief Title: Effect of NT-proBNP Guided Treatment of Chronic Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Netherlands Heart Foundation (Other)
Collaborators: The Interuniversity Cardiology Institute of the Netherlands (Other Government)
Responsible Party: Yigal Pinto, Academic Medical Center, Amsterdam
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2003B131
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2010-02-09 (Estimated); Status verified 2008-08

CONDITIONS: Heart Failure, Congestive
Keywords: NT-proBNP
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NT-proBNP guided treatment group (Active Comparator): In this group, management was guided by an individually set NT-proBNP, defined by the lowest level at discharge or 2 weeks thereafter. If NT-proBNP levels were elevated above the individually set NT-proBNP interventions were performed according to the ESC heart failure guidelines.
  Interventions: Device: NT-proBNP measurements
- Clinically guided arm (Placebo Comparator): Heart failure treatment guided by clinical assessment.
  Interventions: Device: NT-proBNP measurements

INTERVENTIONS:
Device: NT-proBNP measurements

SUMMARY:
The purpose of this study is to determine whether NT-proBNP guided treatment of chronic congestive heart failure will reduce heart failure related morbidity and mortality compared to therapy guided by standard clinical judgement.

ELIGIBILITY:
Inclusion Criteria:

* Admission because of congestive heart failure
* Elevated NT-proBNP levels on admission

Exclusion Criteria:

* Life-threatening cardiac arrhythmias
* Urgent intervention
* Severe lung disease
* Presence of life threatening disease
* Signed informed consent for other study
* Mental or physical status not allowing written informed consent.
* Unwillingness to give informed consent
* Patients undergoing haemodialysis or continuous ambulatory peritoneal dialysis (CAPD)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2004-06; Primary Completion 2009-01 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Difference in total number of days alive and outside the hospital between the NT-proBNP guided and the clinical guided group. | minimum of one year

SECONDARY OUTCOMES:
All cause mortality | at least one year
Cardiovascular mortality | at least one year
All cause hospitalization | at least one year
Cardiovascular related hospitalization | at least one year
Total number of hospitalizations and mortality | at least one year
Total number of cardiovascular hospitalizations and mortality | at least one year
Differences in primary and secondary outcome measures among renal function and age subgroups | At least one year
Differences in evidence based heart failure medication prescription after 3, 6 and 12 months | At least one year
Analysis of major endpoints in patients where NT-proBNP levels were at or below the individual target level in at least 75% of all outpatient visits | at least one year

CONTACTS AND LOCATIONS:
Overall Officials: Dave JW van Kraaij, MD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Universtiy Hospital Maastricht, Maastricht, Limburg, Netherlands

REFERENCES:
- [Derived] Eurlings LW, van Pol PE, Kok WE, van Wijk S, Lodewijks-van der Bolt C, Balk AH, Lok DJ, Crijns HJ, van Kraaij DJ, de Jonge N, Meeder JG, Prins M, Pinto YM. Management of chronic heart failure guided by individual N-terminal pro-B-type natriuretic peptide targets: results of the PRIMA (Can PRo-brain-natriuretic peptide guided therapy of chronic heart failure IMprove heart fAilure morbidity and mortality?) study. J Am Coll Cardiol. 2010 Dec 14;56(25):2090-100. doi: 10.1016/j.jacc.2010.07.030. PMID 21144969
- See also: Interview PRIMA-study ACC congress Orlando 2009 — http://www.acc.org/media/acc_scientific_session_09/press/sunday/ACC09Eurlings_930.pdf